CLINICAL TRIAL: NCT06612424
Title: Comparison of Postoperative Analgesic Efficacy of Quadratus Lumborum Block and Intrathecal Morphine Administration in Cesarean Deliveries
Brief Title: Quadratus Lumborum Block vs Intrathecal Morphine for Post-Cesarean Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, MD, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GaziosmanpasaTREH-ITM
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain
Keywords: intratechal morphine; anterior quadratus lumborum block; cesarean delivery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anterior quadratus lumborum block (Active Comparator): All blocks will be performed by the same anesthesiologist using ultrasound guidance. In the Quadratus Lumborum block group, patients will be placed in the lateral decubitus position. A convex ultrasound probe will be placed in sterile conditions along the midaxillary line, in the subcostal area above the iliac crest, to visualize the quadratus lumborum and psoas major muscles, as well as the L4 vertebral transverse process. Using an in-plane technique, a 22G, 100 mm peripheral block needle will be advanced anterior to the quadratus lumborum muscle and into the subfascial space between the quadratus lumborum and psoas major muscles. After confirming the correct location with hydrodissection, 20 mL of 0.25% bupivacaine will be injected slowly, observing the fascial displacement on ultrasound. The same procedure will be repeated on the contralateral side.
  Interventions: Drug: ANTERİOR QUADRATUS LUMBORUM BLOCK
- intratechal morphine group (Active Comparator): In the intrathecal morphine group, 100 micrograms of morphine (0.1 mL) will be added to the 12 mg of intrathecally administered bupivacaine.
  Interventions: Drug: İNTRATECHAL MORPHİNE GROUP
- control group (No Intervention): Participants in the control group will not receive any interventions such as intrathecal morphine or quadratus lumborum block. They will undergo cesarean sections under spinal anesthesia.

INTERVENTIONS:
Drug: ANTERİOR QUADRATUS LUMBORUM BLOCK — In the Quadratus Lumborum block group, Participants will be placed in the lateral decubitus position. A convex ultrasound probe will be placed in sterile conditions along the midaxillary line, in the subcostal area above the iliac crest, to visualize the quadratus lumborum and psoas major muscles, as well as the L4 vertebral transverse process. Using an in-plane technique, a 22G, 100 mm peripheral block needle will be advanced anterior to the quadratus lumborum muscle and into the subfascial space between the quadratus lumborum and psoas major muscles. After confirming the correct location with hydrodissection, 20 mL of 0.25% bupivacaine will be injected slowly, observing the fascial displacement on ultrasound. The same procedure will be repeated on the contralateral side.
  Arms: anterior quadratus lumborum block
Drug: İNTRATECHAL MORPHİNE GROUP — In the intrathecal morphine group, 100 micrograms of morphine (0.1 mL) will be added to the 12 mg of intrathecally administered bupivacaine.
  Arms: intratechal morphine group

SUMMARY:
İn this study, planned to compare the post-operative analgesic efficacy of Intrathecal Morphine Administration and anterior Quadratus lumborum Block in elective cesarean section operations.

this study primary aim is; To compare the amount of total analgesic use in the first 24 hours in patients

Our secondary aims are: 1.) To compare and evaluate the first rescue analgesia requirement times 2.) To compare the NRS (Numering rating scale) values (resting and dynamic) at 2. 4. 8. 12 . 24. hours in the postoperative follow-up of the patients after anterior Quadratus lumborum block and Intrathecal morphine administration for postoperative analgesia after elective cesarean section operations under spinal anesthesia.

3.) Comparing the side effects such as postoperative nausea and vomiting

DETAILED DESCRIPTION:
Participants scheduled for elective cesarean sections under spinal anesthesia will be divided into three groups: anterior Quadratus Lumborum block (QLB), intrathecal morphine, and control groups, using the sealed-envelope randomization method. All participants will receive detailed information and provide informed consent. Anesthesia for all patients will be administered under spinal anesthesia. Spinal anesthesia will be performed with 12 mg of bupivacaine injected intrathecally at the L3-4 or L4-5 intervertebral space using a 25G spinocan needle.

In the intrathecal morphine group, 100 micrograms of morphine (0.1 mL) will be added to the 12 mg of intrathecally administered bupivacaine. In the QLB and control groups, intrathecal morphine will not be administered, and 0.1 mL of saline will be added to 12 mg of bupivacaine instead. In the anterior QLB block group, the block will be performed postoperatively. Participants in the QLB group will be taken at the end of the surgery.

All blocks will be performed by the same anesthesiologist using ultrasound guidance. In the Quadratus Lumborum block group, participants will be placed in the lateral decubitus position. A convex ultrasound probe will be placed in sterile conditions along the midaxillary line, in the subcostal area above the iliac crest, to visualize the quadratus lumborum and psoas major muscles, as well as the L4 vertebral transverse process. Using an in-plane technique, a 22G, 100 mm peripheral block needle will be advanced anterior to the quadratus lumborum muscle and into the subfascial space between the quadratus lumborum and psoas major muscles. After confirming the correct location with hydrodissection, 20 mL of 0.25% bupivacaine will be injected slowly, observing the fascial displacement on ultrasound. The same procedure will be repeated on the contralateral side. All patients will be monitored in PACU for 30 minutes post-procedure.

The control and intrathecal morphine groups will not receive any postoperative interventions. At the end of the surgery, once the modified Aldrete score is greater than 8, participants will be transferred to the ward due to the spinal anesthesia. Postoperatively, when the spinal anesthesia level recedes by two dermatomes, patients will receive 1g of intravenous paracetamol for analgesia. The postoperative analgesic regimen will include paracetamol 1g every 6 hours (4x1g). In participants with NRS (Numerical Rating Scale) scores greater than 3 during postoperative follow-up, 75 mg of intravenous diclofenac sodium will be administered as rescue analgesia in the ward. Diclofenac was not to be administered more than twice daily, and if the NRS score remained ≥4 despite two doses, intravenous tramadol at a dose of 1 mg/kg was planned.

Participants will be evaluated at 2, 4, 8, 12, and 24 hours postoperatively by a blinded anesthesiologist different from the one who performed the block. Resting and dynamic NRS scores (rated on a scale of 0-10, where 0 indicates no pain and 10 indicates the most severe pain; dynamic NRS scores will be assessed by asking the patient to cough) will be recorded, along with the total amount of analgesics used in the first 24 hours postoperatively, and the incidence of nausea, vomiting, and pruritus will also be evaluated.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

* Participants aged between 18 and 40
* ASA 2 risk group
* Participants at 37-41 weeks of pregnancy
* undergoing cesarean section under spinal anesthesia

Exclusion Criteria:

* The participant does not accept the procedure.
* Patients with a history of eclampsia and preeclampsia during pregnancy
* local anesthetic allergy
* Infection at the procedure site
* Anticoagulant use with bleeding disorder
* Chronic analgesia and opioid use
* Mental, psychiatric and neurological problems -Participant with ASA 3 and above with a history of any chronic disease. -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy women
Enrollment: 118 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
comparing the amount of total analgesic use in the first 24 hours in patients | 24 hour
  For all Participants, postoperative analgesia was planned as paracetamol 1g four times a day for the first 24 hours after surgery. Participants with Numeric Rating Scale (NRS) scores greater than 3 at 2, 4, 8, 12, and 24 hours postoperatively will receive rescue analgesia with diclofenac sodium 75 mg at a dose intravenos.The total diklofenac sodium consumption of participants within the first 24 hours will be compared.
  (At initial trial registration, postoperative NRS pain scores were specified as the primary outcome. During the study phase, total postoperative analgesic consumption was used as the primary outcome for statistical planning, analysis, and reporting.
  The trial registration was updated to ensure consistency between registered outcomes and analyses. NRS pain scores were analyzed as secondary outcomes. This update was not based on study results.)

SECONDARY OUTCOMES:
To compare the NRS (Numering rating scale) values (resting and dynamic) at 2. 4. 8. 12 . 24. hours in the postoperative follow-up of the patients | 24 hour
  To compare the Numeric Rating Scale (NRS) values (at rest and with movement) of the patients during postoperative follow-ups at 2, 4, 8, 12, and 24 hours.Pain intensity was assessed using the Numeric Rating Scale (NRS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores reflect greater pain intensity.
To compare postoperative side effects such as nausea, vomiting, and itching. | 24 hour
  To compare postoperative side effects such as nausea, vomiting, and itching.
time to first rescue analgesic requirement. | 24 hour
  Comparison of the time to first rescue analgesic requirement.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Sehirlioglu, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, 34000, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If requested, it can be provided by contacting the corresponding author.

REFERENCES:
- [Result] Sharpe EE, Molitor RJ, Arendt KW, Torbenson VE, Olsen DA, Johnson RL, Schroeder DR, Jacob AK, Niesen AD, Sviggum HP. Intrathecal Morphine versus Intrathecal Hydromorphone for Analgesia after Cesarean Delivery: A Randomized Clinical Trial. Anesthesiology. 2020 Jun;132(6):1382-1391. doi: 10.1097/ALN.0000000000003283. PMID 32251031
- [Result] Hussain N, Brull R, Weaver T, Zhou M, Essandoh M, Abdallah FW. Postoperative Analgesic Effectiveness of Quadratus Lumborum Block for Cesarean Delivery under Spinal Anesthesia. Anesthesiology. 2021 Jan 1;134(1):72-87. doi: 10.1097/ALN.0000000000003611. PMID 33206131